CLINICAL TRIAL: NCT05249582
Title: The Effect of a Virtual Reality Exergame on Mood
Brief Title: Virtual Reality Compared to Screen Based Engagement on Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto University (Other)
Responsible Party: Principal Investigator, Erick Kim, Ph.D. Doctoral Candidate in Clinical Psychology, Palo Alto University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-075
Record Dates: First submitted 2022-02-01; First posted 2022-02-21 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Virtual Reality
Keywords: virtual reality; mood; technology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Condition (Experimental): Participants will be using a virtual reality headset to engage with a mountain climbing game.
  Interventions: Other: Virtual Reality
- Control Condition (Active Comparator): Participants will be mimicking hand movements displayed on a television screen.
  Interventions: Other: Television Condition

INTERVENTIONS:
Other: Virtual Reality — Virtual reality wireless headset
  Arms: Virtual Reality Condition
Other: Television Condition — Individuals will mimic hand movements of a pre-recorded video of an individual playing the virtual reality climbing game
  Arms: Control Condition

SUMMARY:
Depression has a lifetime prevalence rate of 20.6% and has one of the highest prevalence rates of mental health disorders. Major depressive disorder can lead to higher costs of living for individuals as well as a larger economic decrease associated with inability to work. Current treatment targets one of the two core symptoms of depression of decreased mood or loss of interest in activities. However, current treatment models are not enough because there are more individuals who require treatment than treatment opportunities which creates inequities of care.

Digital interventions provide a unique opportunity to increase widespread accessibility of treatment at reduced and scalable costs. Virtual reality is a newer type of digital intervention that consists of providing experiences for individuals that are different from the physical environment they are currently in. Through audio and visual displays, virtual reality creates a sense of presence, or the experience of immersion, with an environment. Virtual reality has been used in a variety of clinical psychology areas such as training, assessment, and treatment of mental health disorders and other medical conditions. Despite research finding efficacy for virtual reality with anxiety and PTSD, few studies have examined the impact of virtual reality on depressive disorders and low mood. Of studies that have looked at mood changes, most studies measured indirect measures of mood such as energy levels which leads to a gap of research on the efficacy of virtual reality with low mood.

The present study aims to examine if virtual reality exergames improve participant's mood and affect. Additionally, the study will determine if there are different effects of presence, depressive symptoms, and technology familiarity on mood. Furthermore, the study will examine helpfulness and satisfaction to examine usability of virtual reality as a medium for clinical intervention.

DETAILED DESCRIPTION:
Once participants consent, they will complete the three demographic questions and their familiarity with virtual reality. Participants will also complete the Patient Health Questionnaire-8(PHQ-8), Affinity for Technology Interaction scale (ATI), Positive and Negative Affect Schedule (PANAS), and the mood sliding scale. Participants will then be informed that they are going to watch a short clip and press play to watch a 2-minute video of Lion King. After the sad mood induction, participants will complete the PANAS and a mood slider scale. Participants will then be randomly assigned to the virtual reality or control condition. In the virtual reality condition, participants will be asked to complete the first course a virtual reality game called "The Climb". In the control condition, participants will be told that they will be watching a video of a virtual environment climbing game and then be asked to copy all hand movements as accurately as they can. After completing either the virtual reality or control condition, individuals will then complete the PANAS, mood scale, temple presence inventory, three feedback questions, net promoter question, and an open-ended question on improving the activity they just completed. Participants will then be debriefed about the study and compensated for their time.

ELIGIBILITY:
Inclusion Criteria:

* Any individuals who are a general adult population (18-64), be able to read English, and United States Residents. Individuals must be able to read English as all surveys are provided in English.

Exclusion Criteria:

* Individuals who are not part of the general adult population
* Individuals who can not read English
* Individuals who are not United States residents
* Individuals who endorse a history of motion sickness, nausea, migraines, headaches, balance issues, dizziness, epilepsy, neurological conditions where visual stimuli may trigger seizures or other issues, pregnancy, recent concussions, recent illness, recent contagious condition, or other conditions where dizziness, nausea, or headaches are present

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-01-29 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bunge, Ph.D., Principal Investigator — Palo Alto University; Erick Kim, M.S., Principal Investigator — Palo Alto University
Locations (1):
- Palo Alto University, Los Altos, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Virtual Reality Condition | Control Condition
Started | 33 | 31
Completed | 30 | 30
Not Completed | 3 | 1
Not completed — Technical Problems with virtual reality prevented completion | 2 | 0
Not completed — Internet connectivity prevented completion of the condition | 0 | 1
Not completed — Declined to use virtual reality headset | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Reality Condition | Control Condition | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.17 (13.42) | 34.87 (14.52) | 36.02 (13.92)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 13 | 16 | 29
  Female | 15 | 14 | 29
  Not Specified | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0 | 0 | 0
  Asian | 5 | 8 | 13
  Black or African American | 4 | 1 | 5
  Hispanic or Latino | 4 | 7 | 11
  Middle Eastern or North African | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  White | 9 | 12 | 21
  Some Other | 1 | 1 | 2
  No Answer | 1 | 0 | 1
  Multiple | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Positive and Negative Affect Schedule [Mean (Standard Deviation); unit: units on scale] — The Positive and Negative Affect Schedule (PANAS) measures mood through two dimensions: positive affect and negative affect. There are twenty total items of the PANAS and has two subscales that consist of 10 items each on a 5-point Likert scale from 1 (very slightly or not at all) to 5 (extremely). The "moment" instruction was used in the current study to measure current affect. Total scores were reported for each subscale with a range from 10 to 50 for positive affect and 10 to 50 for negative affect. The higher the score for the subscale, the more the individual endorses that affect.
  units on scale
    Positive Affect subscale | 33.83 (8.55) | 30.07 (8.41) | 31.95 (8.62)
    Negative Affect subscale | 14.07 (5.71) | 12.8 (3.84) | 13.43 (4.87)
Mood Sliding Scale [Mean (Standard Deviation); unit: units on scale] — Participant subjective mood rating was measured with a 10-point Likert visual analogue scale from not smiling (1) to smiling (10). Higher scores indicate more positive mood and lower scores indicate more negative mood.
  units on scale | 7.71 (1.54) | 7.6 (1.92) | 7.65 (1.37)

OUTCOME MEASURES:

1. Primary Outcome: Change in Positive Affect and Negative Affect From Baseline to After a 2 Minute Mood Induction
Description: There are twenty total items of the Positive and Negative Affect Schedule. The Positive and Negative Affect Schedule has two subscales, negative affect and positive affect, that consist of 10 items each on a 5-point likert scale from 1 (very slightly or not at all) to 5 (extremely). The PANAS has different time instructions based on when the researcher would like to measure affect and the moment instruction was used. The minimum value for each subscale is 1 and the maximum for each subscale is 5. Each subscale is calculated from an average of 10 items that compose of the subscale. Higher scores indicate more endorsement of positive affect or negative affect depending on the subscale endorsed. Individuals were provided the Positive and Negative Affect Schedule at baseline and after completion 2 minute of mood induction.
Time Frame: Baseline to after 2 minutes of mood induction
Population: Participants in the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Reality Condition | Control Condition
Number analyzed (Participants) | 30 | 30
units on a scale
  Positive Affect Change from Baseline to 2 minute mood induction | 3.7 (7.22) | 4.63 (6)
  Negative Affect Change from Baseline to 2 minute mood induction | 1.97 (3.24) | 1.56 (5.59)

2. Primary Outcome: Change in Positive Affect and Negative Affect From Mood Induction to After Condition Completion
Description: There are twenty total items of the Positive and Negative Affect Schedule. The Positive and Negative Affect Schedule has two subscales, negative affect and positive affect, that consist of 10 items each on a 5-point likert scale from 1 (very slightly or not at all) to 5 (extremely). The PANAS has different time instructions based on when the researcher would like to measure affect and the moment instruction was used. The minimum total value for both positive and negative affect subscales is 10 and the maximum total value for each subscale is 50. Higher scores indicate more endorsement of positive affect or negative affect depending on the subscale endorsed. Participants were measured after mood induction and after completion of the virtual reality or control condition. A change in score was calculated by subtracting the total value of the negative subscale before and after the time point and subtracting the total value of the positive subscale before and after the time point.
Time Frame: Mood induction to after an average of 15 minutes of virtual reality or control condition
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Reality Condition | Control Condition
Number analyzed (Participants) | 30 | 30
units on a scale
  Positive Affect Subscale Change from Mood Induction to After Condition | 8.68 (10.7) | 5.5 (7.3)
  Negative Affect Subscale Change from Mood Induction to After Condition Completion | .21 (5.75) | 2.92 (3.8)

3. Secondary Outcome: Temple Presence Inventory Score Total
Description: The Temple Presence Inventory measures the amount of presence across different technologies such as virtual reality. The Temple Presence Inventory has eight subscales that measure the following dimensions: spatial presence, social presence with actor in medium, passive social presence, active social presence, presence as engagement, presence as social richness, presence as social realism, and presence as perceptual realism. Only spatial presence and presence as engagement was utilized in the study to determine presence as no social interaction was utilized in the study. Each item is rated on a 7-point scale from 1 (not at all) to 7 (very much) with higher mean subscale scores reflecting higher association with the specific presence factor. The minimum value for each subscale was 1 and the maximum value was 7. Each participant was only measured once approximately 30 minutes after the start of study after they completed rather the virtual reality condition or control condition.
Time Frame: One measure after approximately 30 minutes after start of study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Reality Condition | Control Condition
Number analyzed (Participants) | 30 | 30
units on a scale
  Spatial Presence Subscale | 5.71 (.85) | 3.63 (1.64)
  Presence as Engagement subscale | 6.25 (.76) | 3.89 (1.47)

4. Secondary Outcome: Patient Health Questionnaire Depression Scale Total
Description: The Patient Health Questionnaire-8 is an 8-item self-report measure used to screen for major depressive episodes and the severity of depressive symptoms. Each item is rated on a 4-point scale from 0 (not at all) to 3 (nearly every day) with higher mean scores reflecting more depressive symptoms. Individuals were measured once at the beginning of the study. The minimum value for the PHQ-8 was 0 and maximum was 24.
Time Frame: Approximately 5 minutes after start of the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Reality Condition | Control Condition
Number analyzed (Participants) | 30 | 30
units on a scale | 3.21 (3.29) | 4.07 (3.82)

5. Secondary Outcome: Affinity for Technology Interaction Scale Total Score
Description: The Affinity for Technology Interaction Scale is a 9-item measure used to assess an individual's level of engagement with technology. Each item is rated on a 6-point Likert scale from 1 (completely disagree) to 6 (completely agree). Items 3, 6, and 8 are reverse coded and a mean score is calculated with higher scores reflecting an individual having more independence and utilization of technology. Each participant completed the measure once after completion of the virtual reality condition or control condition. The minimum score was 1 and maximum was 6.
Time Frame: Once approximately 30 minutes after start of study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Reality Condition | Control Condition
Number analyzed (Participants) | 30 | 30
units on a scale | 4 (.72) | 3.86 (1.09)

6. Other Pre Specified Outcome: Change in Mood Rating Scale From Baseline to After 2 Minute Mood Induction
Description: Participant subjective mood rating was measured with a 10-point Likert visual analogue scale from not smiling (1) to smiling (10). Higher scores indicate more positive mood and lower scores indicate more negative mood. Minimum score was 1 and maximum was 10. A change in score was calculated by comparing the baseline score to after the 2 minute mood induction.
Time Frame: Baseline to 2 minute mood induction.
Population: Participants in study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Reality Condition | Control Condition
Number analyzed (Participants) | 30 | 30
units on a scale | 1.21 (1.34) | 1.2 (1.06)

7. Other Pre Specified Outcome: Change in Mood Rating Scale
Description: Participant subjective mood rating will be measured with a 10-point Likert visual analogue scale from not smiling to smiling.
Time Frame: Change in affect after average of 15 minutes of virtual reality or control condition
Population: Participants in study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Reality Condition | Control Condition
Number analyzed (Participants) | 30 | 30
units on a scale | 1.76 (1.71) | 1.3 (1.18)

8. Other Pre Specified Outcome: Media Feedback Questions Scores
Description: Participants will be asked three questions on a 7-point Likert scale from 1 (not at all) to 7 (very much) about the difficulty, enjoyment, and helpfulness of the virtual reality or control condition technology. Higher scores indicate more endorsement of difficulty, enjoyment, or helpfulness. Minimum score was 1 and maximum score was 7. Individuals were given the measure once at the end of the study and reported score was utilized with no additional calculations.
Time Frame: Approximately 30 minutes after start of study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Reality Condition | Control Condition
Number analyzed (Participants) | 30 | 30
units on a scale
  Difficulty Question | 4.7 (1.6) | 3.31 (1.52)
  Enjoyment Question | 5.97 (1.45) | 3.79 (1.7)
  Helpfulness Question | 5.4 (1.55) | 3.6 (1.63)

9. Other Pre Specified Outcome: Net Promoter Score
Description: The Net Promoter Score is a single question used to examine an individual's satisfaction with the company or service. Participants answered the question on an 11-point scale from 0 (not likely at all) to 10 (extremely likely), "how likely would you recommend the activity you did to a friend or colleague?". Participants completed the measure at the end of the study with a minimum score of 0 and maximum score of 10. Higher scores represent more endorsement and satisfaction with their experience. Individuals score was reported with no additional calculations.
Time Frame: Approximately 30 minutes after start of study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Reality Condition | Control Condition
Number analyzed (Participants) | 30 | 30
units on a scale | 8.47 (2.2) | 5.49 (3.05)

ADVERSE EVENTS:
Time Frame: Each participant's adverse event data was collected 30-45 minutes after collection of baseline.
Description: No participants reported adverse affects during each session as well as up to the 7 months of study collection date. Before the end of the study, all participants were asked after both virtual reality and control conditions if they were feeling any nausea, dizziness, or other adverse side effects. The total number of individuals at risk was 64, 33 in the virtual reality condition, and 31 in the control condition, and 0 participants endorsed any adverse symptoms.
Arm/Group | Virtual Reality Condition | Control Condition
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/31
Other Adverse Events (participants affected / at risk) | 0/33 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT05249582/Prot_SAP_000.pdf